CLINICAL TRIAL: NCT00001024
Title: A Multicenter, Open-Label Study of Viral Burden in Peripheral Blood Versus Lymphoid Tissue Before and After Antiretroviral Therapy in HIV-Infected Individuals Without AIDS (NOTE: One Arm Receives no Treatment)
Brief Title: The Effects of Anti-HIV Drugs in HIV-Infected Patients Who Do Not Have AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: DATRI 003; 11734 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; AIDS-Related Complex; Zidovudine; Lymph Nodes; Lymphoid Tissue
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
Immunopathogenesis objectives: To compare and quantitatively determine HIV burden and HIV replication in peripheral blood (PB) and lymphoid tissue (LT). To determine the degree to which antiretroviral therapy alters HIV replication in LT.

Clinical objectives: To gain insight into the degree of correlation between immunologic surrogate markers for HIV disease (e.g., CD4, beta-2 microglobulin) as compared to measures of HIV replication in PB and LT. To assess changes in PB and LT viral burden after antiretroviral therapy and to determine its ability to predict an antiviral response.

One of the major problems in defining the immunopathogenic changes in HIV infections has been the inability to correlate the extent of loss of immunologic function with the number of HIV-infected CD4+ cells in the peripheral blood. Few studies exist that measure viral burden in lymph nodes of HIV-infected individuals. Researchers hope to find out whether the amount of HIV virus or markers for the virus in the body's lymph tissue is a better measure of disease progression than the amount of virus or markers for the virus in the blood.

DETAILED DESCRIPTION:
One of the major problems in defining the immunopathogenic changes in HIV infections has been the inability to correlate the extent of loss of immunologic function with the number of HIV-infected CD4+ cells in the peripheral blood. Few studies exist that measure viral burden in lymph nodes of HIV-infected individuals. Researchers hope to find out whether the amount of HIV virus or markers for the virus in the body's lymph tissue is a better measure of disease progression than the amount of virus or markers for the virus in the blood.

Sixteen antiretroviral-naive patients are randomized to either remain antiretroviral-naive (no treatment) or receive zidovudine daily (treatment). Additionally, 16 patients with 26 or more weeks of ongoing zidovudine (AZT) therapy are randomized to either continue on their prestudy AZT regimen or add didanosine (ddI) daily to their baseline AZT dose. Patients remain on their assigned treatment arms for 8 weeks. A lymph node biopsy is performed on day 0 and at week 8. Patients are evaluated at weeks 2, 4, 6, 8 and 9.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis against M. tuberculosis, therapy for oral candidiasis, and short courses (up to 10 days) of acyclovir for herpes lesions.
* Antibiotics as clinically indicated.
* Pneumococcal vaccine and hepatitis B vaccine as medically indicated.
* Regularly prescribed medications such as antipyretics, analgesics, allergy medications, antidepressants, sleep medications, oral contraceptives, or other medications deemed appropriate by the patient's primary care provider.

Recommended:

* PCP prophylaxis if patient's CD4 count falls below 200 cells/mm3 during the study.

Concurrent Treatment:

Allowed:

* Alternative therapies such as vitamins and acupuncture.

Patients must have:

* Documented HIV infection.
* At least two palpable lymph nodes above the waist.
* CD4 counts >= 350 cells/mm3 (if previously antiretroviral-naive) or >= 250 cells/mm3 (if receiving ongoing AZT therapy).

Patients with prior AZT therapy must have received a stable dose of 300-600 mg daily for 26 or more weeks.

Prior Medication:

Required in patients with prior ongoing therapy:

* AZT at dose of 300-600 mg daily for at least 26 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Severe malabsorption.
* Current AIDS-related opportunistic infection, AIDS dementia, AIDS-wasting syndrome, or an AIDS-related malignancy other than minimal Kaposi's sarcoma disease.
* Current medical problems that may interfere with the evaluation of AZT or increase the potential toxicity of AZT (e.g., significant liver disease, diabetes, significant cardiovascular disease, seizure disorders, lymphoma, acute or chronic pancreatitis, or febrile illness).
* Current diagnosis of malignancy for which systemic therapy would be required during study.

Concurrent Medication:

Excluded:

* Ganciclovir, foscarnet, chronic acyclovir, or probenecid.
* Other proven or alleged antiretroviral or anti-HIV drugs.
* Biologic response modifiers.
* Valproic acid.
* Systemic cytotoxic chemotherapy.
* Steroids.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following prior conditions are excluded:

* Prior AIDS-related opportunistic infection, AIDS dementia, AIDS-wasting syndrome, or an AIDS-related malignancy other than minimal Kaposi's sarcoma disease.
* History of medical problems that may interfere with the evaluation of AZT or increase the potential toxicity of AZT (e.g., significant liver disease, diabetes, significant cardiovascular disease, seizure disorders, lymphoma, acute or chronic pancreatitis, or febrile illness).
* History of peripheral neuropathy (patients with prior AZT treatment only).

Prior Medication:

Excluded:

* Prior ddI therapy.
* Less than 26 weeks of prior AZT (in patients with ongoing AZT therapy only).
* Ganciclovir, foscarnet, chronic acyclovir, or probenecid.
* Cytotoxic chemotherapy within 1 month prior to study entry.
* Acute therapy for an infection or other medical illness within 14 days prior to study entry.

History of alcohol abuse (patients with prior AZT treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Cohn, Study Chair; M Niu, Study Chair
Locations (8):
- United States (8):
  - Palo Alto Veterans Affairs Health Care System, Palo Alto, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - Mount Zion Med Ctr / UCSF, San Francisco, California
  - Univ of Illinois, Chicago, Illinois
  - Univ of Maryland at Baltimore, Baltimore, Maryland
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Cohen OJ, Pantaleo G, Graziosi C, Niu M, Fauci AS. Effect of antiretroviral therapy on HIV burden and replication in lymphoid tissue. DATRI 003 Study Group. Int Conf AIDS. 1994 Aug 7-12;10(1):7 (abstract no 001B)